CLINICAL TRIAL: NCT03158688
Title: A Randomized, Open-label, Phase 3 Study Comparing Carfilzomib, Dexamethasone, and Daratumumab to Carfilzomib and Dexamethasone for the Treatment of Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Carfilzomib, Daratumumab and Dexamethasone for Patients With Relapsed and/or Refractory Multiple Myeloma.
Acronym: CANDOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160275; 2016-003554-33 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-18 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Carfilzomib; Dexamethasone; Daratumumab
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; daratumumab; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kd - Carfilzomib and Dexamethasone (Active Comparator): Carfilzomib was administered intravenously (IV) at 20 mg/m^2 in Cycle 1: days 1 and 2; at 56 mg/m^2 in Cycle 1: days 8, 9, 15 and 16. The 56 mg/m^2 dosage was continued in Cycles 2+ on days 1, 2, 8, 9, 15 and 16.
  Dexamethasone was taken by IV infusion at 20 mg on Cycle 1, days 1 and 2 (in Cycles 2+, days 1 and 2 could be either oral or IV) and either orally or by IV infusion on days 8, 9, 15 and 16 and at 40 mg on day 22 of all 28-day cycles.
  Interventions: Drug: Dexamethasone; Drug: Carfilzomib
- KdD - Carfilzomib, Dexamethasone and Daratumumab (Experimental): Carfilzomib was administered intravenously (IV) at 20 mg/m^2 in Cycle 1: days 1 and 2; at 56 mg/m^2 in Cycle 1: days 8, 9, 15 and 16. The 56 mg/m^2 dosage was continued in Cycles 2+ on days 1, 2, 8, 9, 15 and 16.
  Dexamethasone was taken by IV infusion at 20 mg on Cycle 1, days 1 and 2 (in Cycles 2+, days 1 and 2 could be either oral or IV) and either orally or by IV infusion on days 8, 9, 15 and 16 and at 40 mg on day 22 of all 28-day cycles. The administration of dexamethasone was given on carfilzomib and/or daratumumab IV infusion days.
  Daratumumab was administered by IV at 8 mg/kg on Cycle 1: days 1 and 2; at 16 mg/kg on Cycle 1: days 8, 15 and 22, and Cycle 2: days 1, 8, 15, and 22. The 16 mg/kg dosage was continued on Cycles 3-6: days 1 and 15. The 16 mg/kg was further continued on Cycles 7+: day 1 only.
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Carfilzomib

INTERVENTIONS:
Drug: Dexamethasone — Commercially available oral and IV formulas were obtained by investigative sites. Amgen supplied IV or PO dexa for some countries (Poland, Hungry, Romania, Bulgaria, Korea). Dosage modification rules applied based on participant age (participants > 75 years were given lower doses), dexa-related toxicities, and discontinuation of carfilzomib.
Drug: Daratumumab — Daratumumab was supplied as a concentrated solution for infusion in single-use vials.
  Other Names: DARZALEX®
  Arms: KdD - Carfilzomib, Dexamethasone and Daratumumab
Drug: Carfilzomib — Carfilzomib for infusion was supplied as a lyophilized, sterile product in single-use vials. The lyophilized product was reconstituted with preservative-free sterile water for injection, the reconstituted solution contained carfilzomib 2 mg/mL. IV injections lasted approximately 30 minutes.
  Dose could be modified based on a >20% change in body weight or toxicity.
  Other Names: KYPROLIS®

SUMMARY:
Compare carfizomib, dexamethasone, and daratumumab (KdD) to Carfilzomib and dexamethasone (Kd) in terms of progression free survival (PFS) in participants with multiple myeloma who have relapsed after 1 to 3 prior therapies.

DETAILED DESCRIPTION:
This is a phase 3 multicenter, open-label, randomized study in participants with relapsed or refractory multiple myeloma (RRMM) who have received 1 to 3 prior therapies.

Participants receive the treatment determined by randomization for a maximum of approximately 5 years, up to 30 days prior to the final analysis data cutoff (DCO) date or until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or death (whichever occurs first). No crossover between the treatment arms is allowed.

This was an open-label study. However, the assessment of response and disease progression for the primary analysis was determined by an Independent Review Committee (IRC) in a blinded manner. Sensitivity analyses of response and disease progression were determined centrally by the sponsor using a validated computer algorithm (Onyx Response Computational Assessment [ORCA]) in a blinded manner.

Following progression or discontinuation of study drug(s), participants will have 1 follow-up visit (30 days [+3} after last dose of all study drug[s]). After disease progression, data on survival status and subsequent antimyeloma therapy will be gathered at long-term follow-up (LTFU) visits every 12 weeks (+/-2 weeks) until the Final Analysis DCO.

ELIGIBILITY:
Inclusion Criteria:

* Criteria 1 Relapsed or progressive multiple myeloma after last treatment
* Criteria 2 Males or females ≥ 18 years of age
* Criteria 3 Measurable disease with at least 1 of the following assessed within 21 days prior to randomization:
* IgG multiple myeloma: serum monoclonal paraprotein (M-protein) level ≥ 1.0 g/dL,
* IgA, IgD, IgE multiple myeloma: serum M-protein level ≥ 0.5 g/dL,
* urine M-protein ≥ 200 mg/24 hours,
* in subjects without measurable serum or urine M- protein, serum free light chain (SFLC) ≥ 100 mg/L (involved light chain) and an abnormal serum kappa lambda ratio
* Criteria 4 Received at least 1 but not more than 3 prior lines of therapy for multiple myeloma (induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as 1 line of therapy
* Criteria 5 Prior therapy with carfilzomib is allowed as long as the patient had at least a partial response (PR) to most recent therapy with carfilzomib, was not removed due to toxicity, did not relapse within 60 days from discontinuation of carfilzomib, and will have at least a 6-month carfilzomib treatment-free interval from last dose received until first study treatment. (Patients may receive maintenance therapy with drugs that are not proteasome inhibitors or CD38 antibodies during this 6-month carfilzomib treatment free interval)
* Criteria 6 Prior therapy with anti-CD38 antibodies is allowed as long as the patient had at least a PR to most recent therapy with CD38 antibody, was not removed due to toxicity, did not relapse within 60 days from intensive treatment (at least every other week) of CD38 antibody therapy, and will have at least a 6 month CD38 antibody treatment-free interval from last dose received until first study treatment
* Other inclusion criteria may apply

Exclusion Criteria:

* Criteria 1 Waldenström macroglobulinemia
* Criteria 2 Multiple myeloma of IgM subtype
* Criteria 3 POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Criteria 4 Plasma cell leukemia (> 2.0 * 10^9/L circulating plasma cells by standard differential)
* Criteria 5 Myelodysplastic syndrome
* Criteria 6 Known moderate or severe persistent asthma within the past 2 years
* Criteria 7 Known chronic obstructive pulmonary disease (COPD) with a FEV1 < 50% of predicted normal
* Criteria 8 Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, clinically significant electrocardiogram (ECG) abnormalities, screening ECG with corrected QT interval (QTc) of > 470 msec, pericardial disease, or myocardial infarction within 4 months prior to randomization
* Other exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-07-14 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (113):
- United States (11):
  - Lynn Cancer Center Boca Raton Regional Hospital, Lynn Cancer Institute, Boca Raton, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Medical Center - Multiple Myeloma Research Consortium, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Presbyterian Hospital, Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Gabrail Cancer Center, LLC, Dover, Ohio
  - Charleston Oncology, Charleston, South Carolina
  - Baylor Charles A Sammons Cancer Center at Dallas, Dallas, Texas
- Australia (10):
  - Liverpool Hospital, Liverpool, New South Wales
  - St Vincents Hospital Sydney, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Epworth Healthcare, East Melbourne, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, VIC, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
  - Grand HÃ´pital de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
  - Specialized Hospital for Active Treatment of Hematology Diseases EAD, Sofia
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Fakultni nemocnice Plzen, Pilsen
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (8):
  - Centre Hospitalier DÃ©partemental les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier de Versailles - Hopital Andre Mignot, Le Chesnay
  - Centre Hospitalier RÃ©gional Universitaire de Lille - HÃ´pital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers - Hopital la Miletrie, Poitiers
  - Centre Hospitalier Universitaire de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Greece (4):
  - General Hospital Evangelismos, Athens
  - Alexandra Hospital, Athens
  - General University Hospital of Patras Panagia i Voithia, Pátrai
  - Theagenion Cancer Hospital of Thessaloniki, Thessaloniki
- Hungary (5):
  - Bekes Megyei Kozponti Korhaz Dr Rethy Pal Tagkorhaz, Békéscsaba
  - Semmelweis Egyetem, Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Japan (17):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Tesshokai Kameda General Hospital, Kamogawa-shi, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Shibukawa Medical Center, Shibukawa-shi, Gunma
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Medical Center, Kawagoe-shi, Saitama
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Tokushima Prefectural Central Hospital, Tokushima, Tokushima
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
- Poland (6):
  - InterHem, Bialystok
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich w Chorzowie, Chorzów
  - Centrum Onkologii Ziemi Lubelskiej im Swietego Jana z Dukli, Lublin
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im K Marcinkowskiego w Poznaniu, Poznan
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Romania (7):
  - Policlinica de Diagnostic Rapid, Brasov
  - Spitalul Clinic Colentina, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Coltea Clinical Hospital, Bucharest
  - Bucharest Emergency University Hospital, Bucharest
  - Profesor Dr Ion Chiricuta Institut of Oncology, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
- Russia (4):
  - SBHI of Nizhny Novgorod region Regional Clinical Hospital of Nizhny Novgorod na N A Semashko, Nizhny Novgorod
  - SBHI of Republic of Karelia Republic Hosiptal n a V A Baranov, Petrozavodsk
  - State Budget Educational Institution of High Professional Skills Samara State Medical University, Samara
  - Clinic of professional pathology and hematology, Saratov
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (5):
  - Hospital Clinico Universitario de Salamanca, Salamanca, Castilla LeÃ³n
  - Hospital Universitari Germans Trias i Pujol, Badalona, CataluÃ±a
  - Hospital Clinic i Provincial de Barcelona, Barcelona, CataluÃ±a
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Ege University Faculty of Medicine, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
- United Kingdom (3):
  - St James University Hospital, Leeds
  - University College London Hospital, London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Quach H, Nooka A, Samoylova O, Venner CP, Kim K, Facon T, Spencer A, Usmani SZ, Grosicki S, Suzuki K, Delimpasi S, Weisel K, Obreja M, Zahlten-Kumeli A, Mateos MV. Carfilzomib, dexamethasone and daratumumab in relapsed or refractory multiple myeloma: results of the phase III study CANDOR by prior lines of therapy. Br J Haematol. 2021 Aug;194(4):784-788. doi: 10.1111/bjh.17541. Epub 2021 May 28. No abstract available. PMID 34046887
- [Background] Siegel D, Weisel K, Zahlten-Kumeli A, Medhekar R, Ding B, Leleu X. Health-related quality of life outcomes from the CANDOR study in patients with relapsed or refractory multiple myeloma. Leuk Lymphoma. 2021 Dec;62(12):3002-3010. doi: 10.1080/10428194.2021.1941927. Epub 2021 Jun 26. PMID 34180331
- [Background] Suzuki K, Min CK, Kim K, Lee JJ, Shibayama H, Ko PS, Huang SY, Li SS, Ding B, Khurana M, Iida S. Carfilzomib, dexamethasone, and daratumumab in Asian patients with relapsed or refractory multiple myeloma: post hoc subgroup analysis of the phase 3 CANDOR trial. Int J Hematol. 2021 Dec;114(6):653-663. doi: 10.1007/s12185-021-03204-9. Epub 2021 Aug 19. PMID 34410635
- [Background] Usmani SZ, Quach H, Mateos MV, Landgren O, Leleu X, Siegel D, Weisel K, Gavriatopoulou M, Oriol A, Rabin N, Nooka A, Qi M, Beksac M, Jakubowiak A, Ding B, Zahlten-Kumeli A, Yusuf A, Dimopoulos M. Carfilzomib, dexamethasone, and daratumumab versus carfilzomib and dexamethasone for patients with relapsed or refractory multiple myeloma (CANDOR): updated outcomes from a randomised, multicentre, open-label, phase 3 study. Lancet Oncol. 2022 Jan;23(1):65-76. doi: 10.1016/S1470-2045(21)00579-9. Epub 2021 Dec 3. PMID 34871550
- [Background] Landgren O, Weisel K, Rosinol L, Touzeau C, Turgut M, Hajek R, Mollee P, Kim JS, Shu N, Hu X, Li C, Usmani SZ. Subgroup analysis based on cytogenetic risk in patients with relapsed or refractory multiple myeloma in the CANDOR study. Br J Haematol. 2022 Sep;198(6):988-993. doi: 10.1111/bjh.18233. Epub 2022 May 24. PMID 35608261
- [Background] Dimopoulos M, Quach H, Mateos MV, Landgren O, Leleu X, Siegel D, Weisel K, Yang H, Klippel Z, Zahlten-Kumeli A, Usmani SZ. Carfilzomib, dexamethasone, and daratumumab versus carfilzomib and dexamethasone for patients with relapsed or refractory multiple myeloma (CANDOR): results from a randomised, multicentre, open-label, phase 3 study. Lancet. 2020 Jul 18;396(10245):186-197. doi: 10.1016/S0140-6736(20)30734-0. PMID 32682484
- [Background] Leleu X, Beksac M, Chou T, Dimopoulos M, Yoon SS, Prince HM, Pour L, Shelekhova T, Chari A, Khurana M, Zhang J, Obreja M, Qi M, Oriol A, Siegel D. Efficacy and safety of weekly carfilzomib (70 mg/m2), dexamethasone, and daratumumab (KdD70) is comparable to twice-weekly KdD56 while being a more convenient dosing option: a cross-study comparison of the CANDOR and EQUULEUS studies. Leuk Lymphoma. 2021 Feb;62(2):358-367. doi: 10.1080/10428194.2020.1832672. Epub 2020 Oct 28. PMID 33112184
- [Background] Usmani SZ, Quach H, Mateos MV, Landgren O, Leleu X, Siegel D, Weisel K, Shu X, Li C, Dimopoulos M. Final analysis of carfilzomib, dexamethasone, and daratumumab vs carfilzomib and dexamethasone in the CANDOR study. Blood Adv. 2023 Jul 25;7(14):3739-3748. doi: 10.1182/bloodadvances.2023010026. PMID 37163358
- [Background] Weisel K, Mateos MV, Landgren O, Leleu X, Quach H, Bennett L, Talpes M, Majer I, Patel S, Usmani SZ. Health-Related Quality of Life in Patients With Relapsed/Refractory Multiple Myeloma Treated With Carfilzomib, Dexamethasone, and Daratumumab Versus Carfilzomib and Dexamethasone: An Analysis of Patient-Reported Outcomes From the Phase 3 CANDOR Trial. Clin Lymphoma Myeloma Leuk. 2025 Aug;25(8):590-605. doi: 10.1016/j.clml.2025.02.005. Epub 2025 Feb 19. PMID 40087058
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 102 centers. 569 participants were screened and 466 were enrolled. Primary analysis (PA) data cutoff (DCO): 14-Jul-2019. Final analysis (FA) DCO: 15-Apr-2022.
Pre-assignment Details: Participants were randomized in 1:2 ratio to arms KD vs KdD after being stratified by 1) International Staging System (ISS) stage (Stage 1-2 vs Stage 3) at screening, 2) prior proteasome inhibitor exposure (yes/no), 3) number of prior lines of therapy (1 vs ≥ 2), and 4) prior cluster differentiation antigen 38 (CD38) antibody therapy (yes/no).
Groups:
- KdD - Carfilzomib, Dexamethasone and Daratumumab: Carfilzomib was administered intravenously (IV) at 20 mg/m^2 in Cycle 1: days 1 and 2; at 56 mg/m^2 in Cycle 1: days 8, 9, 15 and 16. The 56 mg/m^2 dosage was continued in Cycles 2+ on days 1, 2, 8, 9, 15 and 16.
  Dexamethasone was taken by IV infusion at 20 mg on Cycle 1, days 1 and 2 (in Cycles 2+, days 1 and 2 could be either oral or IV) and either orally or by IV infusion on days 8, 9, 15 and 16 and at 40 mg on day 22 of all 28-day cycles. The administration of dexamethasone was given on carfilzomib and/or daratumumab IV infusion days.
  Daratumumab was administered by IV at 8 mg/kg on Cycle 1: days 1 and 2; at 16 mg/kg on Cycle 1: days 8, 15 and 22, and Cycle 2: days 1, 8, 15, and 22. The 16 mg/kg dosage was continued on Cycles 3-6: days 1 and 15. The 16 mg/kg dosage was continued on Cycles 7+: day 1 only.
Period: Overall Study
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Started | 154 | 312
Treated | 153 | 308
Completed | 49 | 102
Not Completed | 105 | 210
Not completed — Withdrawal by Subject | 14 | 28
Not completed — Decision by sponsor | 13 | 37
Not completed — Lost to Follow-up | 4 | 3
Not completed — Death | 74 | 142

BASELINE CHARACTERISTICS:
Population: Intent to Treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab | Total
Number analyzed (Participants) | 154 | 312 | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.6) | 62.9 (10.0) | 63.4 (9.9)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 77 | 163 | 240
  65 - 74 years | 55 | 121 | 176
  75 - 84 years | 22 | 28 | 50
  >=85 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 135 | 198
  Male | 91 | 177 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 8
  Not Hispanic or Latino | 146 | 291 | 437
  Unknown or Not Reported | 7 | 14 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 46 | 66
  Black or African American | 2 | 7 | 9
  White | 123 | 243 | 366
  Other | 9 | 16 | 25
Frailty Status as Assessed by Investigator [Count of Participants; unit: Participants]
  Fit | 68 | 176 | 244
  Intermediate fitness | 36 | 54 | 90
  Frail | 9 | 10 | 19
  Not available | 37 | 66 | 103
  Missing | 4 | 6 | 10
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    Disease status 0 or 1 | 147 | 295 | 442
    Disease status 2 | 7 | 15 | 22
    Missing | 0 | 2 | 2
Time from Initial Diagnosis to Randomization [Mean (Standard Deviation); unit: months] — Population: Data was not available for some participants.
  months
    number analyzed (Participants) | 149 | 297 | 446
    (all) | 44.03 (36.57) | 47.86 (34.69) | 46.58 (35.34)
Risk Group as Determined by Fluorescent in situ Hybridization (FISH) [Count of Participants; unit: Participants] — The high-risk group consists of the genetic subtypes t(4; 14), t(14; 16), or deletion17p.
  The standard-risk group consists of participants without t(4; 14), t(14; 16), and deletion 17p.
  The unknown risk group is participants with FISH result not done, failed or quantity was not sufficient.
  Participants
    High risk | 26 | 48 | 74
    Standard risk | 56 | 108 | 164
    Unknown | 72 | 156 | 228
Stratification Factor: International Staging System (ISS) Stage per IxRS [Count of Participants; unit: Participants] — The International Staging System (ISS) for myeloma was published by the International Myeloma Working Group (a lower stage indicates less progressed disease):
  Stage I: β2-microglobulin (β2M) < 3.5 mg/L, albumin >= 3.5 g/dL Stage II: β2M < 3.5 mg/L and albumin < 3.5 g/dL; or β2M 3.5 mg/L - 5.5 mg/L irrespective of the serum albumin Stage III: β2M ≥ 5.5 mg/L. Higher stages indicate more advanced disease and/or poorer prognosis.
  Data is the ISS result assessed at the time of randomization using an interactive voice/web response system (IxRS).
  Participants
    Stage I or II | 127 | 252 | 379
    Stage III | 27 | 60 | 87
Stratification Factor: Lines of Prior Treatment per IxRS [Count of Participants; unit: Participants] — Number of participants grouped by total number of prior regimens. Data reported are randomization stratification values.
  Participants
    1 prior treatment | 67 | 133 | 200
    > = 2 prior treatments | 87 | 179 | 266
Stratification Factor: Prior Proteasome Inhibitor Treatment per IxRS [Count of Participants; unit: Participants] — The number of participants with prior proteasome inhibitor treatment assessed at the time of randomization per the IxRS. Data reported are randomization stratification values.
  Participants
    Yes | 139 | 279 | 418
    No | 15 | 33 | 48
Stratification Factor: Prior CD38 Antibody Therapy per IxRS [Count of Participants; unit: Participants] — The number of participants with prior CD38 antibody therapy assessed at the time of randomization per the IxRS. Data reported are randomization stratification values.
  Participants
    Yes | 0 | 1 | 1
    No | 154 | 311 | 465
Geographic Regions [Count of Participants; unit: Participants]
  North America | 12 | 21 | 33
  Europe | 103 | 207 | 310
  Asia Pacific | 39 | 84 | 123

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by the Independent Review Committee (PA DCO Only)
Description: Progression-free survival (PFS) was defined as the time from randomization to the earlier of disease progression or death due to any cause. Participants were evaluated for disease response and progression according to the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC) as assessed by an Independent Review Committee (IRC). The duration of PFS was right censored for participants who met any of the following conditions: 1. no baseline/post-baseline disease assessments; 2. started a new anti myeloma therapy before documentation of progressive disease or death; 3. progressive disease or death immediately after more than 70 days without disease assessment visit or; 4. alive without documentation of disease progression before the analysis trigger date (PA DCO); 5. lost to follow-up or withdrawn consent.
Time Frame: From randomization until the PA DCO date of 14 July 2019; the longest treatment duration as of the DCO was 102.3 weeks
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
Participants
  Participants with PFS events | 68 | 110
  Participants who were censored | 86 | 202
Statistical Analysis 1: Comparison: Kd - Carfilzomib and Dexamethasone vs KdD - Carfilzomib, Dexamethasone and Daratumumab; Stratification factors used in the Log-rank p-value (1-sided) and the Cox model hazard ratio (KdD/Kd) were as assessed at randomization: International Staging System stage at screening (Stage 1 or 2 vs Stage 3); prior proteasome inhibitor exposure (yes vs no); number of prior lines of therapy (1 vs >= 2); Test type: Superiority; p = 0.0014, Log Rank — alpha level of 0.025; Stratified Cox model hazard ratio = 0.630, 95% CI 2-sided [0.464 to 0.854] — KdD/Kd

2. Secondary Outcome: Overall Response (OR) as Assessed by the Independent Review Committee (PA DCO Only)
Description: Overall response rate was defined as the percentage of participants in each treatment group who achieve partial response (PR) or better per the International Myeloma Working Group Uniform Response Criteria (IMWG-URC) as their best response.
  Complete Response (CR): No immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
  Very Good Partial Response (VGPR): Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% reduction in serum M-component with urine M-component <100 mg/24 hours.
  Partial Response (PR): ≥ 50% reduction of serum M-protein and reduction in urine M-protein by ≥ 90% or to < 200 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
  95% CIs for proportions were estimated using the Clopper-Pearson method.
Time Frame: From randomization until the PA DCO date of 14 July 2019; the longest treatment duration as of the DCO was 102.3 weeks
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
percentage of participants | 74.7 [67.0 to 81.3] | 84.3 [79.8 to 88.1]
Statistical Analysis 1: Comparison: Kd - Carfilzomib and Dexamethasone vs KdD - Carfilzomib, Dexamethasone and Daratumumab; Odds ratios and corresponding 95% CIs were estimated using the stratified Mantel-Haenszel method. P-values were calculated using the stratified Cochran-Mantel-Haenszel Chi-Square test; Test type: Superiority; p = 0.0040, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.925, 95% CI 2-sided [1.184 to 3.129] — KdD/Kd

3. Secondary Outcome: Minimal Residual Disease Negative Complete Response Rate (MRD[-]CR) at 12 Months as Assessed by the Independent Review Committee
Description: MRD[-]CR at 12 months was defined as achievement of CR per IMWG-URC by IRC and MRD[-] status as assessed by next-generation sequencing (NGS; at a 10^-5 level) at the 12 months landmark (8 to 13 month window).
Time Frame: 12 Months (8- to 13-month window)
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
percentage of participants | 1.9 [0.4 to 5.6] | 12.8 [9.3 to 17.0]
Statistical Analysis 1: Comparison: Kd - Carfilzomib and Dexamethasone vs KdD - Carfilzomib, Dexamethasone and Daratumumab; Odds ratios and corresponding 95% CIs were estimated using the stratified Mantel-Haenszel method; Test type: Superiority; Odds Ratio (OR) = 7.819, 95% CI 2-sided [2.364 to 25.858] — KdD/Kd

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause. Deaths collected via public source, after end of study were included. Medians were estimated using the Kaplan-Meier method. 95% CIs for medians were estimated using the method by Klein and Moeschberger (1997) with log-log transformation. Participants still alive were censored at the date last known to be alive.
Time Frame: Up to 58 months after the first participant was enrolled (at FA DCO, a median of 40.29 weeks of treatment [any study drug] in the Kd group and 79.29 weeks of treatment [any study drug] in the KdD group; FA DCO was 15 Apr 2022)
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
months | 43.6 [35.3 to NA] — Not enough events to estimate the upper 95% CI | 50.8 [44.7 to NA] — Not enough events to estimate the upper 95% CI
Statistical Analysis 1: Comparison: Kd - Carfilzomib and Dexamethasone vs KdD - Carfilzomib, Dexamethasone and Daratumumab; Hazard ratio and corresponding 95% CIs were estimated using the stratified Cox proportional hazards models. 1-sided p-value from the log-rank test controlling for the randomization stratification factors; Test type: Superiority; p = 0.0417, Log Rank; Cox Proportional Hazard = 0.784, 95% CI 2-sided [0.595 to 1.033] — KdD/Kd

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events are defined as any adverse event with an onset after the administration of the first dose of any study treatment and within the end of study or 30 days of the last dose of any study treatment, whichever occurs earlier.
  The severity of adverse events was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening; Grade 5 = Fatal.
  Treatment-related adverse events are treatment-emergent adverse events considered related to at least one study drug by the investigator, including those with unknown relationship.
Time Frame: PA DCO: the longest treatment duration as of the PA DCO was 102.3 weeks; FA DCO: the longest treatment duration as of the FA DCO was 236.3 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 153 | 308
Participants
  PA DCO: All TEAEs | 147 | 306
  PA DCO: TEAEs: Severity Grade >=3 | 113 | 253
  PA DCO: TEAEs: Serious Adverse Events | 70 | 173
  PA DCO: TEAEs: Leading to discon of carfilzomib | 33 | 65
  PA DCO: TEAEs: Leading to discon of daratumumab | NA — not relevant for this treatment arm | 28
  PA DCO: TEAEs: Leading to discon of dexamethasone | 37 | 33
  PA DCO: Fatal TEAEs | 8 | 30
  PA DCO: Treatment-related TEAEs | 129 | 260
  PA DCO: Related TEAEs: Grade >=3 | 74 | 187
  PA DCO: Related and serious TEAEs | 32 | 84
  PA DCO: Related TEAEs: discon of carfilzomib | 21 | 50
  PA DCO: Related TEAEs: discon of daratumumab | NA — not relevant for this treatment arm | 15
  PA DCO: Related TEAEs: discon of dexamethasone | 24 | 19
  PA DCO: Related Fatal TEAEs | 0 | 5
  FA DCO: All TEAEs | 149 | 306
  FA DCO: TEAEs: Severity Grade >=3 | 120 | 273
  FA DCO: TEAEs: Serious Adverse Events | 80 | 211
  FA DCO: TEAEs: Leading to discontinuation of carfilzomib | 37 | 98
  FA DCO: TEAEs: Leading to discontinuation of daratumumab | NA — not relevant for this treatment arm | 43
  FA DCO: TEAEs: Leading to discon of dexamethasone | 40 | 58
  FA DCO: Fatal TEAEs | 11 | 39
  FA DCO: Treatment-related TEAEs | 131 | 267
  FA DCO: Related TEAEs: Grade >=3 | 82 | 206
  FA DCO: Related and serious TEAEs | 34 | 102
  FA DCO: Related TEAEs: discon of carfilzomib | 22 | 69
  FA DCO: Related TEAEs: discon of daratumumab | NA — not relevant for this treatment arm | 18
  FA DCO: Related TEAEs: discon of dexamethasone | 24 | 30
  FA DCO: Related Fatal TEAEs | 0 | 5

6. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response (DOR) (PA DCO Only)
Description: Duration of response (DOR) was defined as the time (in months) from first evidence of partial response (PR) or better per IMWG-URC by IRC to the earlier of disease progression or death due to any cause for participants with a best response of PR or better. For those who are alive and have not experienced disease progression at the time of data cutoff for analysis, duration of response was right-censored.
  Medians were estimated using the Kaplan-Meier method. 95% CIs for medians were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: From Day 1 until the PA DCO date of 14 July 2019; the longest treatment duration as of the DCO was 102.3 weeks
Population: Participants who responded in the Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 115 | 263
months | 16.6 [13.9 to NA] — Not enough events to estimate the upper 95% CI | NA [NA to NA] — Not enough events to estimate a median and confidence intervals

7. Secondary Outcome: Kaplan-Meier Estimate for Time to Next Treatment (TTNT)
Description: Time to next treatment was defined as the time (in months) from randomization to the initiation of subsequent non-protocol anti-cancer treatment for multiple myeloma. Time to next treatment for participants who do not start the subsequent treatment for multiple myeloma was censored at the date when the participant's information was last available.
  Medians of TTNT duration were estimated using the Kaplan-Meier method. 95% CIs for medians were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: as for outcome 5
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
months
  PA DCO | 17.3 [13.5 to NA] — Not enough events to estimate the upper 95% CI | NA [NA to NA] — Not enough events to estimate a median and confidence intervals
  FA DCO | 17.8 [13.5 to 23.1] | 37.4 [30.1 to 47.8]

8. Secondary Outcome: Kaplan-Meier Estimates for Time to Progression (TTP) as Assessed by the Independent Review Committee (PA DCO Only)
Description: Time to progression was defined as the time (in months) from randomization to documented disease progression. Participants who did not have documented disease progression were censored at the date when data was last available.
Time Frame: From randomization until the PA DCO date of 14 July 2019; the longest treatment duration as of the DCO was 102.3 weeks
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
months | 17.5 [13.2 to NA] — Not enough events to estimate the upper 95% CI | NA [NA to NA] — Not enough events to estimate a median and confidence intervals

9. Secondary Outcome: Time to Progression (TTP): Percentage of Participants Who Had Not Had Disease Progression as Assessed by the Independent Review Committee at Months 3, 6, 12, and 18 (PA DCO Only)
Description: Time to progression was defined as the time (in months) from randomization to documented disease progression. This outcome reports TTP as the percentage of participants who were event free (that is, they had not had disease progression) at the specified time frames. Independent Review Committee assessment for this outcome measure was not planned after the primary analysis.
  95% CIs for event-free rates were estimated using the method by Kalbfleisch and Prentice (1980) with log-log transformation.
Time Frame: Randomization to Months 3, 6, 12, and 18
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
percentage of participants
  3 months | 90.0 [83.7 to 93.9] | 95.3 [92.1 to 97.2]
  6 months | 79.4 [71.6 to 85.3] | 86.4 [81.8 to 89.9]
  12 months | 62.7 [53.6 to 70.5] | 77.5 [72.1 to 82.0]
  18 months | 45.1 [34.5 to 55.4] | 68.5 [62.2 to 74.0]

10. Secondary Outcome: Time to Overall Response as Assessed by the Independent Review Committee (PA DCO Only)
Description: Time to overall response was defined as the time from randomization to the earliest date a response of partial response (PR) or better as per IMWG-URC is first achieved and subsequently confirmed for participants with a best response of PR or better.
Time Frame: From randomization until the PA DCO date of 14 July 2019; the longest treatment duration as of the DCO was 102.3 weeks
Population: Participants who responded in the Intent to Treat Population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 115 | 263
months | 1.5 (1.1) | 1.4 (1.4)

11. Secondary Outcome: Percentage of Participants Who Achieved and Maintained a Minimal Residual Disease Negative Complete Response (MRD[-]CR) for 12 Months or More
Description: A measure of the persistence of the CR (includes strict CR) per International Myeloma Working Group-Uniform Response Criteria (IMWG-URC) and MRD[-] status as assessed by next-generation sequencing (NGS; at a 10^-5 level) for 12 months or more after achieving MRD[-]CR status.
  95% confidence intervals (CIs) for proportions were estimated using the Clopper-Pearson method.
Time Frame: as for outcome 5
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
percentage of participants
  PA DCO | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 1.2]
  FA DCO | 0.0 [0.0 to 2.4] | 5.8 [3.5 to 9.0]

12. Secondary Outcome: Percentage of Participants With a Complete Response (CR) as Assessed by the Independent Review Committee (PA DCO Only)
Description: The percentage of participants in each treatment group who achieved stringent complete response (sCR) or CR per IMWG-URC, as assessed by the IRC, as their best response is presented.
Time Frame: From randomization until the PA DCO date of 14 July 2019; the longest treatment duration as of the DCO was 102.3 weeks
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
percentage of participants | 10.4 [6.1 to 16.3] | 28.5 [23.6 to 33.9]

13. Secondary Outcome: Percentage of Participants Who Achieved Minimal Residual Disease Negative (MRD[-]) Status as Assessed by Next Generation Sequencing at 12 Months
Description: MRD[-] at 12-month was defined as achievement of MRD[-] status as assessed by next-generation sequencing (NGS; at a 10^-5 level) at the 12 months landmark (from 8 months to 13 months window).
  95% confidence intervals (CIs) for proportions were estimated using the Clopper-Pearson method.
Time Frame: 12 Months (8- to 13-month window)
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
percentage of participants | 5.2 [2.3 to 10.0] | 18.3 [14.1 to 23.0]
Statistical Analysis 1: Comparison: Kd - Carfilzomib and Dexamethasone vs KdD - Carfilzomib, Dexamethasone and Daratumumab; Odds ratios and corresponding 95% CIs were estimated by a stratified analysis using the Mantel-Haenszel method; Test type: Superiority; Odds Ratio (OR) = 4.403, 95% CI 2-sided [2.007 to 9.656] — KdD/Kd

14. Secondary Outcome: Quality of Life Core Module (QLQ-C30) Global Health Status/Quality of Life Scores For Baseline Up to the First Follow-Up Visit After the Last Dose
Description: Health-related quality of life was assessed with the use of the European Organization for Research and Treatment of Cancer Quality of Life Core Module (QLQ-C30) questionnaire, a validated instrument in multiple myeloma patients. Scores range from 0 to 100, with higher scores indicating better health related quality of life.
  QLQ-C30 questionnaire was administered prior to dosing every 28 ± 7 days starting from cycle 1 day 1 through first follow-up visit (30 days [+3] after last dose of all study drugs).
Time Frame: Baseline (Day 1 pre-dose) up to 236.3 weeks (longest treatment duration as of the FA DCO)
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
Number analyzed (Participants) | 154 | 312
score on a scale
  Baseline: number analyzed (Participants) | 139 | 289
  Baseline | 66.19 (19.19) | 61.79 (20.37)
  Cycle 2: number analyzed (Participants) | 126 | 281
  Cycle 2 | 64.35 (16.25) | 61.00 (19.65)
  Cycle 3: number analyzed (Participants) | 124 | 264
  Cycle 3 | 66.13 (18.12) | 63.10 (18.24)
  Cycle 4: number analyzed (Participants) | 112 | 258
  Cycle 4 | 66.67 (15.01) | 63.47 (18.66)
  Cycle 5: number analyzed (Participants) | 105 | 252
  Cycle 5 | 67.62 (17.19) | 64.45 (16.76)
  Cycle 6: number analyzed (Participants) | 96 | 244
  Cycle 6 | 68.06 (15.80) | 65.92 (16.85)
  Cycle 7: number analyzed (Participants) | 94 | 223
  Cycle 7 | 69.33 (14.68) | 65.73 (16.59)
  Cycle 8: number analyzed (Participants) | 87 | 206
  Cycle 8 | 69.44 (17.82) | 66.34 (16.64)
  Cycle 9: number analyzed (Participants) | 79 | 202
  Cycle 9 | 65.72 (15.90) | 67.82 (15.53)
  Cycle 10: number analyzed (Participants) | 73 | 197
  Cycle 10 | 68.38 (14.56) | 67.98 (16.26)
  Cycle 11: number analyzed (Participants) | 66 | 189
  Cycle 11 | 67.42 (15.24) | 68.52 (17.37)
  Cycle 12: number analyzed (Participants) | 65 | 187
  Cycle 12 | 65.13 (14.94) | 67.47 (17.16)
  Cycle 13: number analyzed (Participants) | 61 | 175
  Cycle 13 | 67.49 (16.51) | 67.00 (18.21)
  Cycle 14: number analyzed (Participants) | 59 | 169
  Cycle 14 | 67.66 (17.03) | 66.12 (16.60)
  Cycle 15: number analyzed (Participants) | 53 | 167
  Cycle 15 | 69.34 (15.31) | 67.61 (17.68)
  Cycle 16: number analyzed (Participants) | 54 | 165
  Cycle 16 | 68.21 (16.44) | 66.41 (18.69)
  Cycle 17: number analyzed (Participants) | 54 | 159
  Cycle 17 | 69.44 (14.92) | 69.81 (15.28)
  Cycle 18: number analyzed (Participants) | 52 | 155
  Cycle 18 | 66.67 (16.50) | 66.29 (16.38)
  Cycle 19: number analyzed (Participants) | 47 | 150
  Cycle 19 | 69.68 (17.50) | 68.00 (17.33)
  Cycle 20: number analyzed (Participants) | 40 | 141
  Cycle 20 | 71.04 (14.49) | 66.43 (19.52)
  Cycle 21: number analyzed (Participants) | 39 | 143
  Cycle 21 | 70.94 (15.87) | 67.42 (16.25)
  Cycle 22: number analyzed (Participants) | 36 | 139
  Cycle 22 | 68.52 (12.30) | 67.51 (17.90)
  Cycle 23: number analyzed (Participants) | 35 | 131
  Cycle 23 | 69.52 (16.41) | 66.67 (17.63)
  Cycle 24: number analyzed (Participants) | 35 | 125
  Cycle 24 | 68.10 (18.24) | 68.00 (16.51)
  Cycle 25: number analyzed (Participants) | 33 | 127
  Cycle 25 | 67.93 (16.15) | 66.21 (16.78)
  Cycle 26: number analyzed (Participants) | 33 | 121
  Cycle 26 | 70.71 (18.65) | 66.12 (17.54)
  Cycle 27: number analyzed (Participants) | 29 | 112
  Cycle 27 | 65.23 (14.78) | 66.52 (18.35)
  Cycle 28: number analyzed (Participants) | 29 | 109
  Cycle 28 | 63.22 (19.61) | 67.28 (18.66)
  Cycle 29: number analyzed (Participants) | 25 | 105
  Cycle 29 | 66.67 (19.25) | 67.22 (18.10)
  Cycle 30: number analyzed (Participants) | 24 | 104
  Cycle 30 | 67.01 (17.63) | 67.23 (18.52)
  Cycle 31: number analyzed (Participants) | 24 | 101
  Cycle 31 | 68.06 (16.24) | 67.33 (18.81)
  Cycle 32: number analyzed (Participants) | 23 | 94
  Cycle 32 | 66.67 (19.62) | 67.91 (18.45)
  Cycle 33: number analyzed (Participants) | 23 | 91
  Cycle 33 | 67.75 (15.35) | 67.95 (18.92)
  Cycle 34: number analyzed (Participants) | 22 | 86
  Cycle 34 | 68.18 (15.78) | 69.86 (17.77)
  Cycle 35: number analyzed (Participants) | 22 | 88
  Cycle 35 | 65.91 (15.62) | 69.51 (18.00)
  Cycle 36: number analyzed (Participants) | 23 | 86
  Cycle 36 | 63.77 (18.22) | 68.22 (16.93)
  Cycle 37: number analyzed (Participants) | 20 | 89
  Cycle 37 | 67.50 (18.91) | 68.63 (19.01)
  Cycle 38: number analyzed (Participants) | 17 | 84
  Cycle 38 | 65.20 (18.69) | 69.25 (18.47)
  Cycle 39: number analyzed (Participants) | 17 | 78
  Cycle 39 | 64.71 (15.46) | 68.38 (19.15)
  Cycle 40: number analyzed (Participants) | 14 | 78
  Cycle 40 | 58.33 (14.25) | 67.74 (19.34)
  Cycle 41: number analyzed (Participants) | 14 | 79
  Cycle 41 | 66.07 (13.26) | 68.46 (19.37)
  Cycle 42: number analyzed (Participants) | 14 | 68
  Cycle 42 | 63.69 (15.19) | 67.16 (18.77)
  Cycle 43: number analyzed (Participants) | 15 | 57
  Cycle 43 | 67.22 (15.89) | 63.30 (19.91)
  Cycle 44: number analyzed (Participants) | 12 | 50
  Cycle 44 | 61.81 (15.27) | 65.50 (18.21)
  Cycle 45: number analyzed (Participants) | 9 | 41
  Cycle 45 | 67.59 (12.11) | 66.87 (15.53)
  Cycle 46: number analyzed (Participants) | 8 | 34
  Cycle 46 | 64.58 (13.91) | 67.89 (17.66)
  Cycle 47: number analyzed (Participants) | 4 | 27
  Cycle 47 | 66.67 (0.00) | 68.52 (13.74)
  Cycle 48: number analyzed (Participants) | 3 | 22
  Cycle 48 | 61.11 (9.62) | 68.56 (13.35)
  Cycle 49: number analyzed (Participants) | 3 | 19
  Cycle 49 | 61.11 (9.62) | 68.42 (13.49)
  Cycle 50: number analyzed (Participants) | 3 | 16
  Cycle 50 | 61.11 (9.62) | 68.75 (13.09)
  Cycle 51: number analyzed (Participants) | 3 | 12
  Cycle 51 | 63.89 (4.81) | 67.36 (11.49)
  Cycle 52: number analyzed (Participants) | 2 | 9
  Cycle 52 | 54.17 (17.68) | 62.04 (17.24)
  Cycle 53: number analyzed (Participants) | 0 | 3
  Cycle 53 |  | 61.11 (9.62)
  Follow-up: number analyzed (Participants) | 25 | 32
  Follow-up | 61.00 (23.04) | 59.90 (18.02)
Statistical Analysis 1: Comparison: Kd - Carfilzomib and Dexamethasone vs KdD - Carfilzomib, Dexamethasone and Daratumumab; Analysis was performed based on a linear mixed effects model. The model included fixed effects of treatment (all baseline responses were modeled with a dummy treatment), baseline QLQ-C30 GHS/QoL score, randomization stratification factors (ISS stage at screening (Stage 1 or 2 vs Stage 3), prior proteasome inhibitor exposure (yes vs no), number of prior lines of therapy (1 vs ≥ 2)), interaction between treatment and time, and random effects of participant intercept and random slope of time; Test type: Superiority; p = 0.9480, linear mixed effects model; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-2.52 to 2.35], Standard Error of Mean 1.24 — The overall treatment difference (KdD - Kd)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events - any adverse events with an onset after the administration of the first dose of any study treatment and within the end of the study or 30 days of the last dose of any study treatment, whichever occurred earlier. The longest treatment duration as of the FA DCO was 236.3 weeks.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Kd - Carfilzomib and Dexamethasone | KdD - Carfilzomib, Dexamethasone and Daratumumab
All-Cause Mortality (participants affected / at risk) | 80/154 | 148/312
Serious Adverse Events (participants affected / at risk) | 80/153 | 211/308
Other Adverse Events (participants affected / at risk) | 137/153 | 295/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kd - Carfilzomib and Dexamethasone (N=153) | KdD - Carfilzomib, Dexamethasone and Daratumumab (N=308)
Anaemia (Blood and lymphatic system disorders) | 1 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Plasmacytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 4
Angina pectoris (Cardiac disorders) | 2 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 5
Atrial flutter (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 4 | 4
Cardiac failure acute (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 4
Tachycardia (Cardiac disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 3 | 9
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 8
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 3
Hyperthermia (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 14
Sudden death (General disorders) | 0 | 2
Unevaluable event (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Acinetobacter infection (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 6
Campylobacter infection (Infections and infestations) | 1 | 0
Catheter site abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 3 | 14
Lower respiratory tract infection (Infections and infestations) | 1 | 7
Meningitis pneumococcal (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Picornavirus infection (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 16 | 52
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 2
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 2
Pneumonia viral (Infections and infestations) | 2 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 3
Respiratory tract infection (Infections and infestations) | 2 | 8
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 2 | 12
Septic shock (Infections and infestations) | 2 | 5
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 6
Urinary tract infection (Infections and infestations) | 3 | 6
Vascular device infection (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Venous injury (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
C-reactive protein increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Haemoglobin abnormal (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Medical observation (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 8
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 1 | 0
Stupor (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 3
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Hypomania (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 10
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0
Poor venous access (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial enlargement (Cardiac disorders) | 0 | 1
Microvascular coronary artery disease (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 3
COVID-19 pneumonia (Infections and infestations) | 3 | 14
Device related bacteraemia (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Herpes dermatitis (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Dural tear (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Device occlusion (Product Issues) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Hypotonic urinary bladder (Renal and urinary disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dialysis hypotension (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kd - Carfilzomib and Dexamethasone (N=153) | KdD - Carfilzomib, Dexamethasone and Daratumumab (N=308)
Anaemia (Blood and lymphatic system disorders) | 51 | 113
Leukopenia (Blood and lymphatic system disorders) | 6 | 21
Lymphopenia (Blood and lymphatic system disorders) | 13 | 29
Neutropenia (Blood and lymphatic system disorders) | 15 | 49
Thrombocytopenia (Blood and lymphatic system disorders) | 46 | 119
Constipation (Gastrointestinal disorders) | 7 | 23
Diarrhoea (Gastrointestinal disorders) | 27 | 112
Nausea (Gastrointestinal disorders) | 22 | 62
Vomiting (Gastrointestinal disorders) | 13 | 52
Asthenia (General disorders) | 19 | 35
Chills (General disorders) | 7 | 18
Fatigue (General disorders) | 29 | 80
Oedema (General disorders) | 8 | 14
Oedema peripheral (General disorders) | 16 | 38
Pyrexia (General disorders) | 24 | 57
Bronchitis (Infections and infestations) | 21 | 56
Conjunctivitis (Infections and infestations) | 5 | 16
Influenza (Infections and infestations) | 10 | 26
Nasopharyngitis (Infections and infestations) | 15 | 33
Pneumonia (Infections and infestations) | 9 | 38
Respiratory tract infection (Infections and infestations) | 9 | 33
Upper respiratory tract infection (Infections and infestations) | 37 | 104
Urinary tract infection (Infections and infestations) | 3 | 22
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 23
Decreased appetite (Metabolism and nutrition disorders) | 9 | 27
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 29
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 35
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 61
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 41
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 25
Dizziness (Nervous system disorders) | 7 | 24
Headache (Nervous system disorders) | 19 | 47
Neuropathy peripheral (Nervous system disorders) | 6 | 34
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 26
Insomnia (Psychiatric disorders) | 19 | 64
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 55
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 68
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 21
Rash (Skin and subcutaneous tissue disorders) | 10 | 21
Hypertension (Vascular disorders) | 47 | 113
Tachycardia (Cardiac disorders) | 8 | 12
Cataract (Eye disorders) | 11 | 28
Abdominal pain (Gastrointestinal disorders) | 9 | 13
Hypogammaglobulinaemia (Immune system disorders) | 4 | 17
COVID-19 (Infections and infestations) | 3 | 16
Lower respiratory tract infection (Infections and infestations) | 4 | 20
Pharyngitis (Infections and infestations) | 4 | 18
Sinusitis (Infections and infestations) | 5 | 16
Contusion (Injury, poisoning and procedural complications) | 2 | 16
Fall (Injury, poisoning and procedural complications) | 6 | 17
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 19
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 21
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03158688/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03158688/SAP_001.pdf